CLINICAL TRIAL: NCT05685524
Title: Development of Diagnostic Model for Multi-cancer Diagnosis Based on DNA Methylation Biomarkers
Brief Title: Clinical Study of Pan-cancer DNA Methylation Test in Plasma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Wuhan Ammunition Life-tech Co., Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: PanCa
Record Dates: First submitted 2023-01-05; First posted 2023-01-17 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Cancer
Keywords: Colorectal cancer; Liver cancer; Squamous cell carcinoma of the head and neck; Esophageal carcinoma; Pancreatic cancer; Ovarian cancer; Bladder cancer; Cervical cancer; Lung cancer; Stomach cancer
MeSH Terms: conditions — Neoplasms; Colorectal Neoplasms; Liver Neoplasms; Squamous Cell Carcinoma of Head and Neck; Esophageal Neoplasms; Pancreatic Neoplasms; Ovarian Neoplasms; Urinary Bladder Neoplasms; Uterine Cervical Neoplasms; Lung Neoplasms; Stomach Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cancer group: Patients aged 18 years or older with high suspicion of cancer diagnosed by endoscopy, other imaging tests, pathological examinations, etc. The cancer types include liver cancer, head and neck squamous cell carcinoma, esophageal cancer, pancreatic cancer, ovarian cancer, colorectal cancer, bladder cancer, cervical cancer, lung cancer and stomach cancer.
  Interventions: Diagnostic Test: DNA methylation test
- Non-cancer group: Composed by healthy individuals and patients with non-cancerous diseases including hemorrhoids, enteritis, gastritis, tuberculosis and other non-cancerous diseases.
  Interventions: Diagnostic Test: DNA methylation test

INTERVENTIONS:
Diagnostic Test: DNA methylation test — Cell-free DNA were extracted from plasma collected from individuals of cancer and non-cancerous disease groups, then the DNA was bisulfite converted and tested by DNA methylation assay based on real-time PCR platform.

SUMMARY:
We intend to establish an efficient method for plasma cfDNA extraction and Bisulfite transformation to facilitate the detection of DNA methylation status using multiplex fluorescence PCR. Meanwhile, we expect to identify several plasma methylation markers that can be highly sensitive for multi-cancer detection. Finally, we will provide a pan-cancer blood test that is easy to operate, low cost, accurate and easy to promote.

ELIGIBILITY:
Inclusion Criteria:

- (1)age >= 18 years. (2) with high suspicion of cancer diagnosed by endoscopy, other imaging examinations, pathological examinations, etc.

(3) no treatment with radiotherapy or chemotherapy.

Exclusion Criteria:

* (1) received antineoplastic treatment such as radiation/chemotherapy. (2) not preserved as required. (3) contaminated or volume is insufficient. (4) unclear pathological results (5) incomplete patient information.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 200 cases are planned for each cancer type, and the total number of samples in the cancer group is expected to be 2,000.The number of samples in the non-cancer group is expected to be 1000 cases。
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Sensitivity | immediately after the procedure
  The reference standard is the results of histopathological tests
Specificity | immediately after the procedure

CONTACTS AND LOCATIONS:
Locations (1):
- The first affiliated hospital of Zhengzhou University, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yang Q, Dong L, Zhang L, Zhang W, Zhang Y, Huang Y, Jin H, Yang H, Liu X, Zhao Y. Analytical and Diagnostic Performance of a Dual-Target Blood Detection Test for Hepatocellular Carcinoma. Cancer Rep (Hoboken). 2024 Sep;7(9):e70017. doi: 10.1002/cnr2.70017. PMID 39324668